CLINICAL TRIAL: NCT02334956
Title: Linking fMRI to Mobile Technologies in Addiction Research: Pathophysiology of Executive Deficits, Craving and Substance Use
Acronym: MobiCogIm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Fondation pour la Recherche Médicale (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2014/19
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Addiction
Keywords: MRI; Executive Deficits
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient (Experimental): Patient with addiction
  Interventions: Other: Brain MRI
- Control (Experimental): healthy subject
  Interventions: Other: Brain MRI

INTERVENTIONS:
Other: Brain MRI

SUMMARY:
120 individuals with alcohol, cannabis or nicotine dependence as well as healthy controls will be administered a whole-brain imaging exam. The current research project constitutes a highly novel approach to understanding the pathophysiology of addiction through its combination of neuroimaging with state-of-the-art information concerning the real-time expression of risk factors.

DETAILED DESCRIPTION:
* Background : Despite the availability of both pharmacological and psychosocial treatments, most affected individuals will experience addiction as a chronic illness with severe consequences for health outcome. A fundamental challenge to researchers in this domain is therefore to understand the mechanisms leading to relapse. Among the key vulnerability factors associated with addiction chronicity, increasing attention has focused on deficits in executive functions and associated traits (impulsivity, risk taking) that are likely to explain why many individuals with addiction are unable to avoid high-risk contexts or to manage the experience of craving. Research concerning this vulnerability to relapse has been hindered by the manner in which cognitive deficits are traditionally assessed in clinical research. Most commonly, they are thought to represent stable risk factors that show little or no variation within a given individual. However, executive functioning may fluctuate rapidly over time (as does attention, memory, or other key cognitive functions), and therefore comparisons of overall or 'mean' cognitive deficits between healthy and substance-dependent individuals may show no significant differences despite powerful effects of this vulnerability. Therefore, the absence of measurement or characterization of this important relapse mechanism prevents any further research concerning its underlying pathophysiology.
* Purpose : Deficits in executive functioning may explain why many individuals with addiction are unable to avoid high-risk contexts or manage the experience of craving that lead to substance use. The principal objective of this project is to acquire resting state functional Magnetic Resonance Imaging (fMRI) and diffusion tensor imaging (DTI) data on patients with current addiction who will then complete (through a distinct protocol) mobile assessments of daily life executive fluctuations, craving, and substance use.
* Detailed description: 120 individuals with alcohol, cannabis or nicotine dependence as well as healthy controls will be administered a whole-brain imaging exam. The current research project constitutes a highly novel approach to understanding the pathophysiology of addiction through its combination of neuroimaging with state-of-the-art information collected through an independent investigation concerning the real-time expression of risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria patient:
* Aged 18-64 years
* Being affiliated to health insurance
* Having signed an informed consent (later than the day of inclusion and before any examination required by research)
* Participation in the study MOBICOG for patients with addiction
* Fulfils diagnostic criteria for one of the following groups:

Group A: Patients with current (last 12 months) Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) substance addiction (Alcohol / Cannabis / Nicotine); initiation of treatment for addiction within 30 days preceding enrollment in the study; absence of other axis 1 psychiatric disorder currently being treated (by psychotherapy or pharmacotherapy); absence of current or lifetime bipolar disorder or schizophrenia.

Group AM: Patients with current (last 12 months) DSM-IV substance addiction (Alcohol / Cannabis / Nicotine); initiation of treatment for addiction within 30 days preceding enrollment in the study; presence of currently treated unipolar mood disorder (by psychotherapy or pharmacotherapy); absence of current or lifetime bipolar disorder or schizophrenia.

Group AS: Patients currently treated for DSM-IV schizophrenia (last 12 months) with DSM-IV substance addiction (Alcohol / Cannabis / Nicotine); absence of other axis 1 psychiatric disorder currently being treated (by psychotherapy or pharmacotherapy); absence of current or lifetime bipolar disorder.

Inclusion criteria healthy volunteers:

* Aged 18-64 years
* Participation in the study MOBICOG
* Being affiliated to health insurance
* Having signed an informed consent (later than the day of inclusion and before any examination required by research)
* Healthy volunteers without current addiction and with no other currently-treated axis 1 DSM-IV disorder (by psychotherapy or pharmacotherapy); absence of current or lifetime bipolar disorder or schizophrenia

Exclusion Criteria:

* Presence of a counter-indication for MRI
* Presence of any health problem preventing travel to the imaging service of the University Hospital
* Being unable to provide consent to participate
* Pregnant or breastfeeding woman

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Coefficient of correlation between inter-regional hemodynamic signals and clinical and neuropsychological data | After the MRI (D2 at 1 month after the inclusion)

SECONDARY OUTCOMES:
Measurements of daily life functioning through recorded data about craving sensation and executive functioning | After the MRI (D2 at 1 month after the inclusion)
Measurements of brain structure, in relation to brain functioning | After the MRI (D2 at 1 month after the inclusion)

CONTACTS AND LOCATIONS:
Overall Officials: Michèle ALLARD, Prof, Principal Investigator — University Hospital, Bordeaux; Joel SWENDSEN, PhD, Study Director — INCIA-UMR-CNRS 5287
Locations (2):
- France (2):
  - CHU de Bordeaux, Bordeaux
  - Hôpital Charles Perrens, Bordeaux